CLINICAL TRIAL: NCT00299871
Title: A 13-week Multinational, Randomized, Double-Blind, Placebo-Controlled, Dose-Response Trial Assessing the Safety, Tolerability and Efficacy of AVE0010 in Metformin-Treated Subjects With Type 2 Diabetes Mellitus
Brief Title: Dose Ranging Study of the GLP-1 Agonist AVE0010 in Metformin-Treated Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRI6012
Record Dates: First submitted 2006-03-06; First posted 2006-03-07 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lixisenatide

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: LIXISENATIDE (AVE0010)

SUMMARY:
To evaluate the dose-response relationship of AVE0010 administered once daily and twice daily with chronic dosing in metformin-treated subjects with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Males, females, age 30, - 75 years, type 2 diabetes mellitus, treated with metformin ≥1.0 g/day, at a stable dose for at least 3 months, BMI 25 - 40 kg/m2, HbA1C ≥7.0% and <9.0%.

Exclusion Criteria:

* Type 1 diabetes, pregnancy, lactation, women of childbearing potential, treatment with other antidiabetic agents than metformin, history of metabolic acidosis, hemoglobinopathy or hemolytic anemia, clinically significant medical abnormalities.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 542 (Actual)
Dates: Start 2006-02; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
HbA1c levels at baseline and endpoint (at 13 weeks).

SECONDARY OUTCOMES:
Fructosamine, fasting plasma glucose, fasting serum insulin, proinsulin, C-peptide, glucagon.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (7):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Kiev, Ukraine

REFERENCES:
- [Result] Ratner RE, Rosenstock J, Boka G; DRI6012 Study Investigators. Dose-dependent effects of the once-daily GLP-1 receptor agonist lixisenatide in patients with Type 2 diabetes inadequately controlled with metformin: a randomized, double-blind, placebo-controlled trial. Diabet Med. 2010 Sep;27(9):1024-32. doi: 10.1111/j.1464-5491.2010.03020.x. PMID 20722676